CLINICAL TRIAL: NCT02624843
Title: Bioequivalence Study for Benzyl Alcohol Lotion 5% (Hi-Tech Pharmacal Co. LTD) and Ulesfia (Benzyl Alcohol Lotion 5%) (Shionogi Inc.) in the Treatment of Head Lice and Their Ova.
Brief Title: Bioequivalence Study for Benzyl Alcohol Lotion 5%.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akorn, Inc. (Industry)
Collaborators: South Florida Family Health and Research Centers (Network); Axis Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTHP01
Record Dates: First submitted 2015-11-25; First posted 2015-12-09 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Head Lice
MeSH Terms: interventions — Ethanol; Benzyl Alcohols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Benzyl Alcohol Lotion 5% (Experimental): Day 1- Sufficient to saturate hair and scalp for 10 min and then washed out. Day 8 -Sufficient to saturate hair and scalp for 10 min and then washed out.
  Interventions: Drug: Benzyl Alcohol Lotion 5%
- Ulesfia (Benzyl Alcohol Lotion 5%) (Active Comparator): Day 1- Sufficient to saturate hair and scalp for 10 min and then washed out. Day 8 -Sufficient to saturate hair and scalp for 10 min and then washed out.
  Interventions: Drug: Ulesfia (benzyl alcohol lotion) 5%
- Vehicle Placebo Lotion 0% (Placebo Comparator): Day 1- Sufficient to saturate hair and scalp for 10 min and then washed out. Day 8 -Sufficient to saturate hair and scalp for 10 min and then washed out.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benzyl Alcohol Lotion 5% — White topical lotion
  Arms: Benzyl Alcohol Lotion 5%
Drug: Ulesfia (benzyl alcohol lotion) 5% — White topical lotion
  Arms: Ulesfia (Benzyl Alcohol Lotion 5%)
Drug: Placebo — White topical lotion
  Arms: Vehicle Placebo Lotion 0%

SUMMARY:
To establish the therapeutic equivalence and safety of a generic Benzyl Alcohol Lotion 5% with Ulesfia Lotion 5% in eradication of head lice in the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant females aged 6 month or over with an upper age limit of 60 years.
* Prospective participants upon examination are confirmed to have at least 3 live head lice (defined as lice adults or nymphs) and at least 5 viable appearance louse eggs (nits).
* Prospective participants who give written informed consent or, if the participant is under 17 years of age, whose parent/guardian gives written informed consent to participate in the study.
* Prospective participants who will be available for follow up visits over the 21 days following first treatment.
* Prospective female participants (including female caregivers) of childbearing potential who are willing to provide a urine pregnancy test.
* Prospective participants who agree not to shave their hair or use any other pediculicide, nit combing, or louse treatment method during the course of the study.

Exclusion Criteria:

* Prospective participants with a known sensitivity to any of the ingredients in benzyl alcohol lotion 5% (Hi-Tech Pharmacal Inc) or Ulesfia 5% (Shionogi Inc).
* Prospective participants with a known history of irritation or sensitivity to pediculicides or hair care products.
* Prospective participants with a secondary bacterial infection of the scalp (eg. impetigo/pyoderma) or have a secondary or long term scalp condition that could make it difficult to evaluate the extent and severity of an infestation or that would present a problem in the evaluation of response to therapy (e.g., psoriatic lesions of the scalp, extensive seborrheic dermatitis).
* Prospective participants who have been treated with other head lice products within 4 weeks prior to randomization.
* Prospective participants who regularly shave their hair, have bleached their hair, used a permanent color on their hair, or their hair has been permanently straightened or waved within the previous 2 weeks.
* Prospective participants who have been treated with Trimethoprim containing products within the previous 4 weeks, or who are currently taking such a course.
* Females who are pregnant, planning to become pregnant, during the course of the study period, or are currently breast feeding mothers.
* Females of childbearing potential who are unwilling to use an adequate method of contraception from at least 4 weeks prior to the first application of treatment and until 4 weeks after the last application of treatment, or who are unwilling to take a urine pregnancy test.
* Prospective participants who have participated in another clinical study or used an investigational new drug within 1 month before entry into this study.
* Participants who have already participated in this clinical study.

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 239 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Rivera, Principal Investigator — South Florida Family Health and Research Centers; Lydie Hazan, MD, Principal Investigator — Axis Clinical Trials; Patrick Clarke, MD, Principal Investigator — Axis Clinical Trials; Lidia E Serrano, Principal Investigator — South Florida Family Health and Research Centers; Nancy Pyram-Bernard, D.O., Principal Investigator — South Florida Family Health and Research Centers; Ian F Burgess, M.Phil., Study Director — Insect Research and Development LTD
Locations (3):
- United States (3):
  - Axis Clinical Trials, Los Angeles, California
  - South Florida Family Health and Research Centers (Lice Source Services Inc), Miami, Florida
  - South Florida Family Health and Research Centers (Lice Source Services Inc), Plantation, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Benzyl Alcohol Lotion 5% | Ulesfia (Benzyl Alcohol Lotion 5%) | Vehicle Placebo Lotion 0%
Started | 107 | 108 | 24
Completed | 70 | 72 | 16
Not Completed | 37 | 36 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzyl Alcohol Lotion 5% | Ulesfia (Benzyl Alcohol Lotion 5%) | Vehicle Placebo Lotion 0% | Total
Number analyzed (Participants) | 107 | 108 | 24 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 77 | 85 | 18 | 180
  Between 18 and 65 years | 30 | 23 | 6 | 59
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 98 | 24 | 224
  Male | 5 | 10 | 0 | 15
Region of Enrollment [Number; unit: participants]
  United States | 107 | 108 | 24 | 239

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infestation Successfully Eliminated by Active Treatment.
Description: Successful elimination of infestation by active treatment [Time frame: 22 + 2 days]. No evidence of active head lice infestation 22 days after enrollment.
Time Frame: Study Day 22 +/-2
Population: PP
Measure: Count of Participants; unit: Participants
Arm/Group | Benzyl Alcohol Lotion 5% | Ulesfia (Benzyl Alcohol Lotion 5%) | Vehicle Placebo Lotion 0%
Number analyzed (Participants) | 70 | 72 | 16
Participants | 59 | 57 | 6

ADVERSE EVENTS:
Arm/Group | Benzyl Alcohol Lotion 5% | Ulesfia (Benzyl Alcohol Lotion 5%) | Vehicle Placebo Lotion 0%
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/108 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/108 | 0/24
Other Adverse Events (participants affected / at risk) | 2/107 | 1/108 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzyl Alcohol Lotion 5% (N=107) | Ulesfia (Benzyl Alcohol Lotion 5%) (N=108) | Vehicle Placebo Lotion 0% (N=24)
Skin, nervous system and general disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Hot paraesthesia on scalp
redness of eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — redness of eyes
fever (General disorders) | 0 (0) | 1 (1) | 0 (0) — fever

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No